CLINICAL TRIAL: NCT04073043
Title: A Pilot Randomized Trial of a Telephone Coaching Intervention for Postpartum Depression and Anxiety
Brief Title: Telephone Coaching Intervention for Postpartum Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Jane McCusker, MD DrPH, Principal Scientist, St. Mary's Research Centre, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMHC-18-25
Record Dates: First submitted 2019-04-17; First posted 2019-08-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Depression; Anxiety
Keywords: Support; Self-management; Resources
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The intervention is a secure psychoeducational e-health platform. Participants will be randomized into two groups - Intervention and Control and will be provided with access to self-guided learning modules such as emotional health, healthy living, mental fitness tools and parenting. The Intervention group will also be given telephone coaching by a trained lay coach who will guide participants through the materials, provide positive reinforcement and help to answer questions. The coach will schedule 7 contacts over the 12 week intervention period with an average of 10 - 15 minutes for each call. A suggested script with specific objectives is provided as well as training based on the drafted coach manual. Coach supervision meetings will take place where difficulties/questions will be reviewed including coach logs, recorded contacts periodically and feedback to the coach. The control group will be provided with the intervention materials but will not receive telephone support.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will have access to the web-based intervention along with telephone coaching. Participants in the intervention will receive 7 coach calls over a period of 12 weeks.
  Interventions: Behavioral: Telephone Coaching
- Control Group (No Intervention): The control group will have access only to the web-based intervention without telephone support

INTERVENTIONS:
Behavioral: Telephone Coaching — Access to Telephone Coaching for a period of 12 weeks
  Arms: Intervention Group

SUMMARY:
Mental health problems affect up to 20% of women at some point during the perinatal period (i.e., from pregnancy to one year postpartum. Perinatal mental health (PMH) problems have been associated with many negative obstetric outcomes, such as higher elective caesarean section, premature delivery, pre-eclampsia, lower fertility rates, and longer postpartum hospital stay.

This research study is a pilot randomized controlled trial (RCT) to assess the feasibility, acceptability, and potential benefits of a low cost sustainable web-based intervention (WBI) with telephone coaching for women with mild to moderate symptomatology of postpartum depression and anxiety.

The intervention contains modules that will help postpartum mothers:

1. Learning new information to better understand their condition. This can help mothers feel that they are not alone, and that their experience is not abnormal. It gives a better understanding that can help them feel more confident in their communications with health care professionals and can make it easier to share their experience with family and friends.
2. Learning and practicing new skills. This can help mothers feel confident that they can engage in the behaviours that have been shown to be beneficial for mood and to improve stress. This can include learning to plan activities like physical exercise, practice proper sleep hygiene or learning to use a new way of thinking about problems to help you find solutions.

This trial represents a first step to implement a sustainable intervention for PMH problems in order to better serve women's PMH needs and preferences for support. This will help inform the current gap in low cost web-based interventions for PMH.Specific deliverables (in both French and English) include: a manual detailing coaching procedures; reports for decision makers and short summaries for stakeholder groups

DETAILED DESCRIPTION:
Among women who present with symptoms of depression or anxiety within 5 - 12 weeks of giving birth, the following research questions will be considered:

1. Feasibility and Acceptability of the two intervention components - WBI and coaching:

   a) Among women in the coached and non-coached groups: i) What are participant perceptions of the usability of the WBI with regard to the layout, navigation and functionality at 3 months following randomization? ii) What are the rates of satisfaction with the intervention at 6 months? b) Among women in the coached group: i) What are rates of completion of the planned telephone contacts? ii) What are participant perceptions of the acceptability of the coaching at 6 months? iii) What are coach perceptions of acceptability of coaching intervention?
2. Effectiveness: The EPDS is the primary outcome measure for depression and the GAD-7 is the primary outcome measure for anxiety i) Primary outcomes: What is the effect of coaching on the severity of depression and/or anxiety symptoms at the 3 and 6 month follow-up? ii). Secondary outcomes: What is the effect of coaching at 3 and 6 months on maternal functioning, parental stress and at 6 months on use of mental health services, and barriers to use of these services?

Hypothesis: The investigators expect a decrease in scores in the EPDS and GAD-7 in the group with coaching when compared to the group without coaching at 6 months.

The investigators will conduct a pilot single -blind randomized control trial with lay telephone coaching with two groups of women, one assigned to the WBI with coaching and the other to the self-guided WBI. This RCT would consist of the following steps:

1. Recruiting a sample of women immediately post-birth(24 hrs) at SMHC and obtaining consent to contact them again within 5 - 12 weeks postpartum
2. 5-12 weeks postpartum: Screen women for eligibility for RCT;
3. Request informed consent to RCT
4. Baseline measures (T0);
5. Follow up at 3 months (T1) and
6. Follow-up at 6 months (T2). Women who deliver elsewhere in the CIUSSS can be referred to the study at 5-12 weeks postpartum. These women then follow steps 2-6

The participants will be asked to answer online questionnaires at each time point as mentioned above and use web-based resources for information and support after giving birth. The intervention group will receive telephone support from coaches to help answer questions and navigate the website material.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ (at birth)
* Ability to speak English or French
* Livebirth
* Access to the internet and email

Inclusion criteria (at step 2):

* Score on either EPDS 10 - 19 or GAD-7 of 10+. Women with a GAD-7 score of 15+ will be referred to the mental health nurse and will be included in the study.
* Baby at home

Exclusion Criteria:

* Women currently undergoing psychological treatment and /or having a history of bipolar disorder or psychosis will be excluded
* Severe symptoms (Score of 20 or more on the EPDS, will be excluded Any anti-depressant and/or psychological treatment will be managed by the participant's own physician and not by the research team.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Screening, 3 months & 6 months
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure, with a four point response scale, and is designed to screen participants for depressive symptoms in the last seven days. The EPDS includes one question (Item 10) about thoughts of self-harm. Sum scores for the 10 items are used to generate a total score. This measure has optimal sensitivity and specificity using a cut-off score of 12. For the purposes of this study, a cut off score of 10+ is used to identify participants with potentially clinically significant depressive symptoms . Women who score 20 or over on the EPDS will be excluded and is considered to be in the range of severe symptoms. A score of 10-19 will be included in the study and is considered to be mild to moderate symptoms. An increase in these scores in either category would be consdiered as an increase in symptoms of depression
Generalized Anxiety Disorder-7 (GAD-7) | Screening,3 months & 6 months
  The seven-item, self-report Generalized Anxiety Disorder (GAD-7) questionnaire, designed to screen for and measure the level of anxiety symptoms during the last seven days. An identified cut point of 10 is used for this study. Women who have a GAD-7 of greater than 15 will be considered as showing symptoms of anxiety in the severe range. a score of 10 - 15 will be considered mild to moderate symptoms of anxiety.

SECONDARY OUTCOMES:
Questions on usability & acceptability | 3 months
  All participants will complete a survey at 3 months after randomization to assess usability (layout, navigation, functionality) and acceptability (overall usefulness, usefulness of specific topics, utility of the site for improving mood and engaging in healthy behaviours, credibility and program length/duration). System usage data will complement users' self-reports and include frequency and duration of user log in, number of modules viewed. Given that a mean adherence rate of about 50% (defined as number of modules completed) has been observed in e-mental health interventions showing significant changes in outcomes, this cut-off has been selected as an acceptable usage metric.
Barkin Index of Maternal Functioning (BIMF) | Baseline, 3 months & 6 months
  The Barkin Index of Maternal Functioning (BIMF) is designed to measure maternal functioning in new mothers. It is known for its comprehensibility, patient-centered assessment style, and psychometric profile. The 20 item BIMF is based on the experiences of women experiencing new motherhood and has a possible range of 0 to 120 with a total score of 120 indicating optimal maternal functioning.
Parental Stress Questionnaire (PARSS) | Baseline, 3 months & 6 months
  The Parental Stress Questionnaire (PARSS) is an 18 item questionnaire designed to measure the positive aspects of parenting as well as the negative stressful aspects. The self-report five point scale helps parents rate how they feel about the relationship with their child by agreeing or disagreeing on various themes of parenting. The tool is used to assess the change in level of stress and would inform the level of support or services need to improve parenting capacity. The 8 positive items are reverse scored so that possible scores on the scale can range between 18-90. Higher scores on the scale indicate greater stress.
Client Satisfaction Questionnaire (CSQ-8) | 6 months
  Satisfaction with the intervention will be measured with an 8-item open-ended questions that will ask participants what they liked most about the intervention and what could be improved.
Questionnaire on Use of services for mental health problems | Baseline & 6 months
  This measure uses questions adapted from the Canadian Community Mental Health Questionnaire (CCMHS). These questions ask about visits to psychiatrists, psychologists, family doctors, nurse, social workers, self-help groups, and other community services for mental health problems since they entered the study. The questions will identify the percentage of women who have used these services since the time they entered the study.
Acceptability of Coaching Questionnaire | 6 months
  The intervention group will receive an additional questionnaire at 6 months on the usefulness (positive and negative aspects) of having support and guidance from the coach
Coach logs and records | 6 months
  Adherence to the coaching will be tracked in coach logs that record attempted and completed, duration of contacts, topics covered, modules that were recommended and/or used, goals set, and problems that arose. Contacts will be tape-recorded for fidelity monitoring.
Coach exit interview | 6 months
  At the end of the study, the coach will participate in a semi structured exit interview regarding their experiences, the challenges that arose in delivering this form of support, and how the intervention could be improved.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Schwartz, MDCM, Principal Investigator — McGill University
Locations (1):
- St. Mary's Hospital Centre, Montreal, Quebec, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT04073043/Prot_SAP_000.pdf